CLINICAL TRIAL: NCT07362316
Title: Longitudinal Evaluation of Neuromuscular Involvement in Type 1 Myotonic Dystrophy
Acronym: NatHis DM1
Status: Completed | Type: Observational
Sponsor: Institut de Myologie, France (Other)
Responsible Party: Sponsor
Other Study IDs: NatHis DM1
Record Dates: First submitted 2026-01-14; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Steinert Myotonic Dystrophy
Keywords: Steinert Myotonic Dystrophy; DM1; Natural history
MeSH Terms: conditions — Myotonic Dystrophy | interventions — Dental Occlusion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DM1 patients: Adults, no intervention
  Interventions: Other: Quantification of myotonia; Other: MyoAnkle; Other: Measurement of exercise-induced fatigue; Other: Moviplate; Other: 6-minute walk test; Other: Test du Box and Blocks; Other: Purdue board test; Other: 9-hole test; Other: Balance measurement
- Healthy controls: Adults, no intervention
  Interventions: Other: Quantification of myotonia; Other: MyoAnkle; Other: Measurement of exercise-induced fatigue; Other: Moviplate; Other: 6-minute walk test; Other: Test du Box and Blocks; Other: Purdue board test; Other: 9-hole test; Other: Balance measurement

INTERVENTIONS:
Other: Quantification of myotonia — Measurement of relaxation time after exertion
Other: MyoAnkle — Measurement of ankle flexion and extension strength
Other: Measurement of exercise-induced fatigue — Measurement of exercise-induced fatigue
Other: Moviplate — Measurement of movement coordination and fatigue
Other: 6-minute walk test — The subject must walk between two cones separated by 25 m. During this test, a measurement of the quality of the walk will also be carried out using an accelerometer.
Other: Test du Box and Blocks — Measures gross manual dexterity
Other: Purdue board test — assessment of finger dexterity and gross hand, finger and arm movements
Other: 9-hole test — Evaluation of motor skills and coordination of the upper limbs
Other: Balance measurement — Balance measurement on a force platform

SUMMARY:
Primary objective: To determine the sensitivity to change of neuromuscular functional outcomes during the natural (non-interventional) progression of myotonic dystrophy type 1 (DM1), in order to identify the most relevant and robust outcome measures for use in therapeutic trials.

Secondary objective: To compare patients with DM1 to healthy control subjects to assess the discriminative power of biomechanical and electrophysiological parameters.

Study design: This is an open-label, single-center observational study with no direct individual benefit.

Participants: Thirty patients with DM1 will be evaluated three times over a three-year period, while thirty control subjects will be assessed once.

Timeline: The planned inclusion period is 12 months, with a follow-up duration of 36 months, resulting in a total study duration of 48 months.

Functional assessment-particularly muscle strength-is essential for both diagnosis and longitudinal monitoring of neuromuscular diseases. In therapeutic trials, outcome measures must meet strict scientific requirements, including precision, sensitivity, and reliability. Muscle strength is frequently used as a primary or secondary endpoint in trials targeting neuromuscular disorders. Even modest functional improvements resulting from therapy must be detectable with sensitive measurement tools.

Myotonic dystrophy is the most common muscular dystrophy in adults, with an estimated prevalence of 1 in 8,000. It is a genetic disorder inherited in an autosomal dominant manner. Two genetically distinct forms are recognized: myotonic dystrophy type 1 (DM1, or Steinert disease) and the rarer, more recently identified type 2 (DM2). This study focuses on DM1 due to its higher prevalence and greater clinical severity.

The study will assess parameters related to myotonia, muscle strength, motor function, and neuromuscular excitability. Patients will be evaluated every 18 months over a three-year period. Control subjects will undergo a single assessment. The expected outcome is the identification of the most robust and sensitive parameters for longitudinal monitoring of DM1 patients, particularly in the context of future therapeutic trials.

A similar study will be conducted in parallel in Quebec (Principal Investigator: Prof. Jack Pumirat, CHU de Québec). Data common to both centers will be analyzed jointly.

DETAILED DESCRIPTION:
Background and Rationale Assessment of functional capacities-particularly muscle strength-is essential for both diagnosis and follow-up of patients with neuromuscular diseases. In therapeutic trials, measurement tools must meet strict scientific requirements: accuracy, sensitivity, and reliability. Muscle strength is frequently used as a primary or secondary outcome in clinical trials. Even small functional improvements must be detectable to demonstrate therapeutic benefit.

Myotonic dystrophy is the most common adult muscular dystrophy (prevalence ~1/8,000). It is an autosomal dominant genetic disorder with two distinct forms: type 1 (DM1, Steinert disease) and type 2 (DM2), the latter being rarer. This study focuses on DM1 because of its higher prevalence and more severe clinical manifestations.

More than a century after its first description, DM1 remains highly complex. It shows extreme clinical variability in:

* Age of onset (from congenital or prenatal forms to late-onset after age 60),
* Severity (from asymptomatic to severe neonatal forms),
* Initial organ involvement (heart, central nervous system, skeletal muscle, eye, etc.).

Marked intrafamilial variability is also observed.

Muscular manifestations include:

1. Myotonia, mainly affecting the hands, characterized by delayed muscle relaxation.
2. Progressive muscle weakness and atrophy, predominantly affecting distal muscles of the limbs, face, and neck.

Despite advances in molecular understanding and preclinical therapies, validated, sensitive, and reproducible tools for longitudinal clinical assessment-especially muscle function-remain limited. Knowledge of the natural history of DM1 is incomplete, and few studies have used highly sensitive functional outcome measures.

Current Assessment Methods and Limitations

Muscle function is commonly evaluated using:

* Manual Muscle Testing (MMT, MRC scale),
* Quantitative Muscle Testing (QMT) with dynamometers,
* Timed functional scales. MMT is simple and widely used but suffers from low sensitivity and poor reproducibility. Large sample sizes are required to detect small changes. QMT provides numerical data suitable for statistical analysis but remains evaluator-dependent and insufficiently sensitive in DM1. Prior studies suggest muscle function declines by approximately 1-3% per year in DM1, highlighting the need for more sensitive tools, especially for trials with limited patient numbers.

New Measurement Devices and Study Purpose Highly sensitive ergometers (e.g., MyoGrip, Myo-Ankle) have been developed to assess very weak patients. These devices have been technically validated, with established normative data and standardized procedures.

This study aims to validate these tools in adult DM1 patients and to improve understanding of disease progression. It is part of an international research program supporting gene therapy development and validation of reliable, non-invasive clinical outcome measures.

Study Design

* Type: Monocentric, open-label, non-interventional study
* Duration: 3 years of follow-up (total study duration: 48 months)
* Participants:

  * 30 genetically confirmed adult DM1 patients
  * 30 age- and sex-matched healthy controls
* Assessment points:

  * Patients: baseline, 18 months, 36 months
  * Controls: baseline only
* A parallel protocol is conducted in Québec (Canada). Study Objectives Primary Objective To determine the sensitivity to change of neuromuscular functional outcomes during the natural progression of DM1, in order to select the most relevant endpoints for therapeutic trials.

Secondary Objective To compare DM1 patients with healthy controls to assess the discriminative power of biomechanical and electrophysiological measures.

Outcome Measures

The study includes a comprehensive battery of assessments:

1. Myotonia Quantification

   * MyoTone Test: measures force relaxation times after voluntary contraction.
   * Provides sensitive indicators such as half-relaxation time and relaxation slope.
2. Ankle Strength Measurement

   * Isometric dorsiflexion and plantarflexion using the Myo-Ankle ergometer.
   * Complemented by manual dynamometry and MMT.
3. Strength of Selected Muscle Groups

   o Eight representative muscle groups measured with a handheld dynamometer (IMADA).
4. Exercise-Induced Fatigability

   * Standardized sustained contraction at 60% maximal force.
   * Combined force measurements, nerve stimulation, and high-density surface EMG using Laplacian electrodes.
   * Non-invasive and suitable for longitudinal follow-up.
5. Moviplate Test

   o Measures rapid alternating wrist and finger movements over 30 seconds.
6. 6-Minute Walk Test

   * Conducted according to international guidelines.
   * Gait quality assessed with an accelerometer (Locometrix).
   * Followed by a 30-second normal-speed walking test.
7. Upper Limb Functional Tests

   * Box and Blocks Test
   * Purdue Pegboard Test
   * 9-Hole Peg Test
8. Balance Assessment

   o Postural control measured on a force platform under four sensory conditions.
9. Additional Data Collected

   * Demographics, anthropometrics, body composition
   * Clinical scales (MIRS)
   * Quality of life (INQoL)
   * Disability (Rotterdam Handicap Scale) Statistical Analysis

Data will be anonymized and analyzed using SPSS and Statview. Analyses include:

* Descriptive statistics,
* Sensitivity to change (Standardized Response Means),
* Repeated-measures ANOVA for longitudinal changes,
* Correlations with clinical and functional parameters,
* Joint analysis with the Canadian center, including center effects. Ethical and Regulatory Aspects
* Conducted according to French law, Good Clinical Practice, the Declaration of Helsinki, and data protection regulations.
* Approved by an ethics committee (CPP) and relevant authorities.
* Written informed consent required.
* No expected individual benefit and no financial compensation.
* Risks are minimal and limited to transient muscle discomfort.
* Data confidentiality strictly maintained.
* Documents archived for 15 years. Expected Impact

Although no direct benefit is expected for participants, this study aims to:

* Validate highly sensitive, reliable outcome measures,
* Improve knowledge of the natural progression of DM1,
* Facilitate future therapeutic trials, including gene therapy, in small patient populations.

ELIGIBILITY:
Inclusion Criteria:

For patients:

* Diagnosed with myotonic dystrophy type 1 confirmed by genetic analysis
* Presenting with motor weakness (MIRS score of 3 or 4)
* Able to walk for ten minutes
* Able to be informed and provide informed consent
* Affiliated with a French social security scheme

For healthy subjects:

* Matched in age (± 1 year) and sex to patients
* Able to be informed and provide informed consent
* Affiliated with a French social security scheme

Exclusion Criteria:

* for patients and control subjects
* Participation in another ongoing biomedical research study
* Orthopaedic disorders of the ankle or hand
* Epilepsy
* Progressive cancer
* Insulin-dependent diabetes
* Uncontrolled heart disease, congestive heart failure, uncontrolled heart rhythm disorders (supraventricular or ventricular) or severe cardiac conduction disorders (AVB II or III or HV > 70 ms) without pacemaker (patients with pacemakers may be included) [echocardiography within one year prior to inclusion]
* Unstabilised and uncontrolled hypertension under treatment (or treated with Propranolol, Prazosin or Clonidine) or blood pressure greater than 160/90 mmHg in the supine position
* Dementia syndrome, major depressive disorder
* History of drug or alcohol abuse in the last six months
* Vital capacity < 50% or total lung capacity < 50%, daytime mechanical ventilation (EFR less than 2 years old)
* Hypercapnia (PaCO2 ≥ 8 Kpa or 60 mmHg) (blood gas less than 2 years old)
* Visual disorders incompatible with the performance of the tests (e.g. cataracts, etc.)
* Women who are pregnant, breastfeeding or not using effective contraception
* Patients treated with cyclosporine
* Any condition that, in the investigator's opinion, would be incompatible with the proper conduct of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients will be recruited during neurological consultations at hospitals participating in the study. Healthy subjects will be recruited either from among the patients' friends and family members who are known not to carry the mutation, or through announcements made during consultations.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-09-23 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2015-12-15 (Actual)

PRIMARY OUTCOMES:
Determine sensitivity to changes in neuromuscular functional criteria | 18 and 36 months after baseline
  Determine sensitivity to changes in neuromuscular functional criteria during the natural progression (non-interventional follow-up) of patients with myotonic dystrophy type 1 in order to select the most relevant follow-up criteria during a therapeutic trial.

SECONDARY OUTCOMES:
Comparison of variables from patients with myotonic dystrophy type 1 and control subjects | Baseline
  Compare a population of patients with myotonic dystrophy type 1 with a population of control subjects to determine the discriminatory power of biomechanical and electrophysiological criteria.

CONTACTS AND LOCATIONS:
Locations (2):
- Centre de recherche du CHU de Québec-Université Laval, Laval, Canada
- Institut de Myologie, Paris, Île-de-France Region, France